CLINICAL TRIAL: NCT00403182
Title: The CORE Study (Chemotherapy OR Endocrine Treatment First?) A Randomized Study by the Scandinavian Breast Group [CORE]
Brief Title: Chemotherapy and Hormone Therapy as First-Line Therapy in Treating Postmenopausal Women With Metastatic or Locally Advanced Breast Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: study halted prematurely, prior to enrollment of first participant
Sponsor: Technical University of Munich (Other)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000515936; KRDI-TUM-CORE-GYN-040-380-2126; EU-20660; EUDRACT-2005-000986-20; KRDI-TUM-COR-259-PAE-0100-I
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy; Letrozole

INTERVENTIONS:
Drug: chemotherapy
Drug: letrozole

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by lowering the amount of estrogen the body makes. It is not yet known whether giving chemotherapy before hormone therapy is more effective than giving hormone therapy before chemotherapy in treating breast cancer.

PURPOSE: This randomized phase III trial is studying chemotherapy to see how well it works when given before or after hormone therapy as first-line therapy in treating postmenopausal women with metastatic or locally advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the optimal sequence of chemotherapy and endocrine therapy as first-line therapy in postmenopausal women with metastatic or locally advanced breast cancer that is potentially sensitive to both modalities.

OUTLINE: This is an open-label, randomized, crossover, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I (chemotherapy first): Beginning within 4 weeks after randomization, patients receive chemotherapy* comprising either an anthracycline- or a taxane-based regimen, or a combination of both drugs, according to local institutional guidelines. Treatment continues for 6 months or longer, in the absence of disease progression or unacceptable toxicity. After discontinuation of chemotherapy, patients receive endocrine therapy comprising oral letrozole once daily in the absence of disease progression or unacceptable toxicity. Patients with immediately life-threatening disease (e.g., lymphangitis carcinomatosa or liver involvement exceeding 1/3 of the liver) are recommended for second-line chemotherapy.

NOTE: *Patients may receive chemotherapy on a separate clinical chemotherapy trial but must first undergo randomization in this study.

* Arm II (endocrine therapy first):Beginning immediately after randomization, patients receive oral letrozole once daily in the absence of disease progression or unacceptable toxicity. Patients who demonstrate progressive disease then receive chemotherapy as in arm I.

Quality of life and pain are assessed at baseline and then periodically for 5 years.

After completion of study therapy, patients are followed periodically.

PROJECTED ACCRUAL: A total of 1,500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Metastatic or locally advanced disease
  * Bilateral breast cancer allowed
* Measurable or evaluable progressing metastases or local disease

  * No sclerotic bone metastases as only disease
  * Measurable or evaluable disease not in a previously irradiated area
* No immediately life-threatening metastatic disease
* No known HER2/neu positivity, as defined by either of the following:

  * 3+ by immunohistochemistry
  * HER2-positive by fluorescent in situ hybridization or chromogenic in situ hybridization
* No known cerebral or leptomeningeal metastases
* Hormone receptor status:

  * Estrogen and/or progesterone receptor positive tumor

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal, as defined by any of the following:

  * Bilateral oophorectomy and amenorrhea > 3 months
  * Radiation castration and amenorrhea > 3 months
  * Spontaneous menopause and amenorrhea > 12 months
  * Previous hysterectomy and age > 55 years
* ECOG performance status 0-2

  * Must be ambulant with organ function and performance status adequate for conventional combination chemotherapy
* No serious hypersensitivity to letrozole or other components of study drug
* No other prior or concurrent malignancy except for basal cell carcinoma or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* No prior systemic treatment for recurrent or metastatic breast cancer
* No other concurrent radiotherapy, endocrine therapy, cytotoxic therapy, or experimental therapy for cancer

Max Age: 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Response to first and second treatment modalities as assessed by RECIST criteria
Time to first and second progression
Toxicity and safety as assessed by NCI CTCAE v3.0
Quality of life as assessed by Hospital Anxiety and Depression Scale (HADS-D), Functional Assessment of Cancer Therapy-General (FACT-G), FBK-R23, and FLZ-G periodically for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Paepke, MD, Study Chair — Technical University of Munich
Locations (9):
- Germany (9):
  - Kreiskrankenhaus, Ebersberg
  - Gynaekologische Gemeinschaftspraxis - Pause, Thiel & Neuhofer, Freising
  - Frauenklinik Universitaet Giessen, Giessen
  - Klinikum Ingolstadt, Ingolstadt
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Munich Oncologic Practice at Elisenhof, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Praxis Kowolik Prechtl-Sattler, Munich
  - Abt. Innere Medizin Onkologic, Schwarzenberg